CLINICAL TRIAL: NCT02578160
Title: Efficacy of Tell-Show-Do Behavior-Management Technique in Anxiety, Pain and Behavior Levels During an Inferior Alveolar and Lingual Nerve Block Procedure in Preschool Children: A Randomized Clinical Trial
Brief Title: Efficacy of Tell-Show-Do Behavior-Management Technique During Local Anesthesia in Preschool Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Evelyn Alvarez Vidigal (Other)
Responsible Party: Sponsor-Investigator, Evelyn Alvarez Vidigal, PhD Student, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBEMATECH
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Dental Anxiety; Pain; Infant Behavior; Heart Rate and Rhythm Disorders
Keywords: pain; infant behaviour; heart rate; dental anxiety
MeSH Terms: conditions — Pain; Infant Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tell-Show-Do Behavior Technique (Experimental): This technique will involve verbal explanations related to the inferior alveolar and lingual nerve block procedure in phrases appropriate to the developmental level of the patient (tell);demonstrations for the patient of the visual, auditory, olfactory, and tactile aspects of the procedure in a carefully defined, nonthreatening setting (show); and then, without deviating from the explanation and demonstration, completion of the procedure (do).
  Interventions: Procedure: inferior alveolar and lingual nerve block procedure
- "Conventional Technique" (Active Comparator): The operator will explain how he/she will do the inferior alveolar and lingual nerve block procedure in phrases appropriates to the child. Then quietly cover the child's field of view by hand during the inferior alveolar and lingual nerve block.
  Interventions: Procedure: inferior alveolar and lingual nerve block procedure

INTERVENTIONS:
Procedure: inferior alveolar and lingual nerve block procedure — inferior alveolar and lingual nerve block

SUMMARY:
This will be a randomized, controlled, parallel-group clinical trial. The aim of this study will be to evaluate the effectiveness of "Tell-Show-Do" Behavior Management Technique versus a Conventional technique (covering the patient's vision) during an inferior alveolar and lingual nerve block in preschool children referred for treatment at the School of Dentistry, University of Sao Paulo, Brazil. The sample will consist of 52 children from 3 years old to 5 years 11 months old who need dental pulp treatment and / or tooth extraction of primary molars. Preschool children with no history of allergies to Lidocaine anesthetic or systemic/neurological diseases and who did not take local anesthesia before the study will be include in this research.

DETAILED DESCRIPTION:
Children will be randomly allocated to treatment groups (n = 26 for each group) according to the technique: (1) Tell-Show-Do and (2) Conventional. Anxiety and pain will be evaluated by the scale of Facial Image (EIF) and Wong-Baker Pain Scale, respectively. The cooperation of the patient will be evaluated by behavioral scale Frankl.

ELIGIBILITY:
Inclusion Criteria:

1. Preschool children with severe dental caries who need dental pulp treatment and / or tooth extraction of inferior primary molars.

Exclusion Criteria:

1. Preschool children with history of allergies to Lidocaine (local anesthetic)
2. Preschool children with systemic or neurological diseases
3. Preschool children who have received local dental anaesthesia before this study

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Preschool children's anxiety levels changes before and after anesthesia procedure - Facial Image Scale (FIS) | Baseline and after one week
  The children will be asked to point at which face they felt most like at that moment (row of five faces ranging from very happy to very unhappy - FIS)

SECONDARY OUTCOMES:
Preschool children's pain levels - Wong-Baker FACES Pain Scale | At the end of the local anesthesia procedure (2 minutes)
  The children were asked to point at which face they felt most like at that moment (row of six faces ranging from very happy-does not hurt to very unhappy-hurt as much as you can imagine)
Preschool children's behavior - Frankl Behavioral Rating Scale | Baseline and during the local anesthesia procedure (2 minutes)
  It will be evaluated children's behavior (definitely negative, negative, definitely positive, positive) during de local anesthesia procedure
Heart rates | Baseline and during local anesthesia procedure
Parent's anxiety levels - Corah's dental anxiety scale (DAS) - parent questionnaire | Baseline
family socioeconomic indicators - questionnaire related to socioeconomic conditions | Baseline
  questionnaire related to family socioeconomic conditions

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Bönecker, Study Director — University of Sao Paulo
Locations (1):
- Faculdade de Odontologia da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
July 2016